CLINICAL TRIAL: NCT06346483
Title: Comparison of Ureteroscopy With High-powered Holmium:Yag Laser Lithotripsy With and Without Moses 2.0 Pulse Modulation
Brief Title: Ureteroscopy With High-powered Holmium:Yag Laser Lithotripsy With and Moses On or Moses Off
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Professor of Urology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00218929
Record Dates: First submitted 2024-03-22; First posted 2024-04-04 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Kidney Stone; Ureteral Stone
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis | interventions — Dust

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moses 2.0 arm (Active Comparator): Ureteroscopy with high powered holmium laser lithotripsy with Moses 2.0 pulse modulation.
  Ureteral dusting settings: 0.2-0.3x60 Hz (not to exceed 20 W) Renal dusting settings: 0.2-0.3 J x 120 Hz (not to exceed 40 W)
  Interventions: Procedure: Dusting with Moses 2.0 Modulation; Other: Moses 2.0 Modulation
- Standard High-powered arm (Active Comparator): Ureteroscopy with high powered holmium laser lithotripsy without Moses 2.0 pulse modulation.
  Ureteral dusting settings: 0.2-0.3 x 60 Hz (not to exceed 20 W) Renal dusting settings: 0.2-0.5 J x 80 Hz standard (not to exceed 40 W)
  Interventions: Procedure: Dusting without Moses 2.0 Modulation

INTERVENTIONS:
Procedure: Dusting without Moses 2.0 Modulation — Dusting is when a laser is used to break a stone down into tiny fragments that are able to pass through the urine.
  Arms: Standard High-powered arm
Procedure: Dusting with Moses 2.0 Modulation — Dusting is when a laser is used to break a stone down into tiny fragments that are able to pass through the urine.
  Arms: Moses 2.0 arm
Other: Moses 2.0 Modulation — Lumenis Pulse™ 120H Holmium Laser System with MOSES™ 2.0 Technology used for lithotripsy and BPH treatments
  Arms: Moses 2.0 arm

SUMMARY:
The purpose of this study is to compare Moses 2.0 pulse modulation technology and the standard high powered Holmium Laser lithotripsy and how it will affect time in the operating room, time using the laser, laser energy, and stone free rates.

Currently Moses 2.0 laser technology is FDA approved and currently used in practice since 2021. No study to this date has compared Moses 2.0 without pulse modulation laser technology to Moses 2.0 with pulse modulation laser technology.

The study will be including kidney and ureteral stones (a kidney stone located in the tube between the kidney and the bladder) that are 6mm and greater, but less than 20 mm in size undergoing ureteroscopic treatment. High powered lasers are used for "dusting". Dusting is when a laser is used to break a stone down into tiny fragments that are able to pass through the urine.

DETAILED DESCRIPTION:
On the day of surgery, the treatment assigned to the patient will be determined by chance, like flipping a coin. Neither the patient nor the study doctor will choose the treatment type. Each patient will have an equal chance of being given either surgical treatment. One group will have stones treated with high powered laser dusting with Moses 2.0 pulse modulation and the dust produced will pass spontaneously through the urine. The other group will have stones treated with standard of care high power laser fragmentation and the dust produced will pass spontaneously through the urine. The surgical procedure will not differ from the treatment a patient would receive if he/she were not in this study.

8 to 12 weeks after surgery, participants will undergo a standard of care renal bladder ultrasound (RBUS) and Kidney Ureter Bladder Abdominal X-ray (KUB) to evaluate for stones and hydronephrosis, which is swelling of the kidney due to build-up of urine.

If there are abnormal findings on the RBUS or KUM at the 8 to 12 week follow-up, participants will be asked to return to the urology clinic and may have to repeat imaging to ensure participants did not develop a postoperative condition.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ureteroscopy and laser lithotripsy
* Stone size ≥8 but < 20 mm in the proximal ureter or kidney. Multiple stones ≤4 are allowed. Bilateral surgeries are allowed
* Willing to sign informed consent

Exclusion Criteria:

* Staged surgery
* Nephrocalcinosis
* Participant is less than 18 years of age
* Inability to provide informed consent
* Members of vulnerable patient populations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-09-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Operative time | Day of procedure
  Total amount of time (in minutes) taken to complete the procedure.
Stone Free Rate | 6-8 weeks post procedure
  This is measured by KUB and Renal bladder ultrasound that is post-operative standard of care.
  Stone free is defined as no stone fragments seen on KUB or RBUS. If there are hyperechoic fragments seen on RBUS but not KUB and the stone analysis was not uric acid, the patient will be considered stone free. The investigators will also calculate a clinically stone free rate (< 4mm residual fragments allowed).
  The Stone Free Rate assessments by the investigators will highlight the rate, or ratio of patients who are stone free and patients who are not stone free after procedure.

SECONDARY OUTCOMES:
Lasing time | Day of procedure
  (no residents, fellows will be allowed under attending supervision)
Total laser energy (kJ) | Day of procedure
  The energy setting of the laser that is used during procedure.
Detection of postoperative strictures | 12 weeks
  If postoperative ultrasound shows hydronephrosis at follow up. Repeat Ultrasound will be obtained 1 month later. If hydronephrosis persists, CT urogram will be obtained. If stricture is identified, then appropriate intervention will be recommended.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Krambeck, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States